CLINICAL TRIAL: NCT05244148
Title: A Multicentre, Randomised, Open Label, Parallel Group, Controlled Clinical Trial to Evaluate Efficacy and Tolerability of Two Seawater-based Formulations Plus a Standard of Care Versus the Standard of Care Alone for Relief of Nasal Congestion in Paediatric Subjects With Common Cold
Brief Title: Two Seawater-based Formulations for Relief of Nasal Congestion in Paediatric Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit 300 subjects.
Sponsor: Church & Dwight Company, Inc. (Industry)
Collaborators: Evidilya S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST-20-F11
Record Dates: First submitted 2022-01-03; First posted 2022-02-17 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Common Cold; Nasal Congestion
Keywords: Common Cold; Nasal Congestion; Children
MeSH Terms: conditions — Common Cold; Nasal Obstruction | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 3 Arms:
  1. Group A: IP1 - Stérimar BLOCKED NOSE Baby nasal spray + standard of care
  2. Group B: IP2 - Stérimar Stop & Protect Cold Baby + standard of care
  3. Group C: Standard of Care alone
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): IP1 - Stérimar BLOCKED NOSE Baby nasal spray + standard of care
  Interventions: Device: IP1 - Stérimar BLOCKED NOSE Baby nasal spray; Behavioral: Standard of Care
- Group B (Experimental): IP2 - Stérimar Stop & Protect Cold Baby + standard of care
  Interventions: Device: IP2 - Stérimar Stop & Protect Cold Baby + standard of care; Behavioral: Standard of Care
- Group C (Other): Standard of Care alone
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Device: IP1 - Stérimar BLOCKED NOSE Baby nasal spray — 1 to 2 sprays per nostril at least 2 twice a day and, as needed, up to a maximum of 6 times a day.
  Arms: Group A
Device: IP2 - Stérimar Stop & Protect Cold Baby + standard of care — 1 to 2 sprays per nostril at least 2 twice a day and, as needed, up to a maximum of 6 times a day.
  Arms: Group B
Behavioral: Standard of Care — hydration + rest at home + if needed paracetamol

SUMMARY:
The objective of this clinical trial is to evaluate the tolerance and efficacy of two Stérimar nasal sprays products in children who have nasal congestion due to the common cold.

DETAILED DESCRIPTION:
This clinical trial is a multicentre, randomized, parallel-group, controlled, open-label clinical trial to evaluate the efficacy of two Stérimar nasal sprays formulations (medical device already CE marked) for nasal congestion in children aged 3 to 48 months with common cold. In total the study foresees 300 patients divided between the different clinical sites.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female infants and toddlers aged 3 - 48 months (inclusive) at enrolment (Day 0).
2. Caretaker(s) answering "yes" to the question "Do you feel that your child has a cold?" at enrolment (Day 0).
3. Subjects with symptoms started within 48 hours prior to enrolment (Day 0).
4. Subjects with nasal congestion (blocked / stuffy nose) rated as at least grade 2 (moderately bothersome) on a 0 to 2-point scale, based on morning evaluation (within an hour of subject awakening).
5. Subjects showing at least grade 2 on a 0 to 2-point scale for at least one of the following additional signs of cold symptoms: runny nose, nasal crust (dry mucus), thick mucus, sneezing and cough.
6. Legal caretaker(s) signed written informed consent for their young ones to participate in the study.
7. Legal caretaker(s) willing to comply with all study procedures.
8. Ability of the caretaker(s) (in the Investigator's opinion) to comprehend the full nature, procedures, and purpose of the study.

Exclusion Criteria:

1. Subjects presenting a body temperature greater than 38°C measured with a non-contact infrared thermometer at enrolment (Day 0).
2. Subjects presenting any secondary infection (such as bronchitis, otitis, tracheitis, pneumonia, and so on) at enrolment (Day 0).
3. Subjects with positive results on a streptococcal antigen screening test (rapid antigen detection test or RADT) at enrolment (Day 0).
4. Subjects with history of allergic rhinitis.
5. Subjects presenting any congenital or chronic disease that in the opinion of the Investigator would adversely affect the results of the study (e.g., asthma, pneumonia, laryngotracheobronchitis, sinusitis, and so on).
6. Subjects presenting any kind of immunodeficiency.
7. Subjects presenting any hypersensitivity or allergy or intolerance to any component of the study products.
8. Subjects with a positive medical history to any significant illness within the 2 weeks prior to the enrolment (Day 0).
9. Subjects presenting any active systemic infection or medical condition that may require treatment or therapeutic intervention during the study.
10. Subjects currently participating or having participated in another clinical trial during the last 30 days prior to enrolment (Day 0).
11. Subjects using saline nose drops or nasal sprays or pumps other than the study products, antibiotics, antivirals, intranasal medicines, decongestants, antihistamines, echinacea, combination cold formulas, supplements containing ≥ 10 mg zinc that would influence symptoms scores at enrolment (Day 0) within 12 hours prior the day of screening.

Ages: 3 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Change of nasal congestion. | Through study completion, an average of 10 days
  Assess change of nasal congestion, evaluated by means of a specific questionnaire ("Cold Symptom Severity" questionnaire), to be completed at Day 0 (baseline) and daily from the beginning to the end of the study; comparisons among groups A, B versus group C.

SECONDARY OUTCOMES:
Change of other cold symptoms. | Through study completion, an average of 10 days
  Assess change of other cold symptoms, evaluated by means of a specific questionnaire ("Cold Symptom Severity" questionnaire), to be completed at Day 0 (baseline) and daily from the beginning to the end of the study; comparisons among groups; comparisons among groups A, B versus group C.
  Other cold symptoms:
  * Nasal crust (dry mucus)
  * Runny nose (drip/sniff/snorting/drainage/discharge)
  * Thick mucus
  * Sneezing
  * Cough.
Occurrence of secondary infections. | Daily through the end of the study, approximately 10 days
  Assessment of occurrence of secondary infections (number) daily, from the beginning to the end of the study; comparisons of group A, B versus group C. Secondary infections will be confirmed by the Investigator.

OTHER OUTCOMES:
Onset of relief. | Through study completion, an average of 10 days
  Assessment of onset of relief (immediate relief) after the entire product application is completed (1 or 2 sprays) at Day 0 (baseline) and daily from Day 1 to Day 3 of the study; comparisons within groups A and B.
Concomitant medications. | Through study completion, an average of 10 days
  Assessment of use of concomitant medications (frequency, excluding paracetamol) will be done from the beginning to the end of the study; comparisons among groups A, B, C.
Frequency of paracetamol administration. | Through study completion, an average of 10 days
  Assessment of use of paracetamol (frequency) will be done from the beginning to the end of the study; comparisons within groups A, B, versus group C.
Quality of sleep. | Through study completion, an average of 10 days
  Assessment of quality of sleep will be evaluated by means of the "quality of sleep" questionnaire, to be completed at Day 0 (baseline) and daily from the beginning to the end of the study; comparisons within groups A, B versus group C.
Global assessment on common cold status. | Through study completion, an average of 10 days
  Global assessment on common cold status will be evaluated by means of the "global assessment on common cold status" questionnaire, to be completed from the beginning to the end of the study; comparisons within groups.

CONTACTS AND LOCATIONS:
Locations (1):
- San Paolo Hospital, Milan, Italy